CLINICAL TRIAL: NCT02007174
Title: Triple Subconjunctival Bevacizumab Injection for Early Recurrent Pterygium. One Year Follow-up
Brief Title: Bevacizumab Injection for Recurrent Pterygium
Status: Completed | Type: Observational
Sponsor: Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Sponsor
Other Study IDs: CC-002-2011
Record Dates: First submitted 2013-12-02; First posted 2013-12-10 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Recurrent Pterygium
Keywords: recurrent pterygium; bevacizumab; triple dose
MeSH Terms: conditions — Pterygium | interventions — Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Bevacizumab injection: Three subconjunctival intralesional injections of bevacizumab. Bevacizumab injections were 2.5 mg/0.05 ml, subconjunctivally applied near to the pterygium recurrence. Application of bevacizumab was performed three times: basal, 2 and 4 weeks.
  Interventions: Drug: Bevacizumab
- Medical Treatment: In order to reduce the patient bias, the control eye received a sham laser treatment, under slit lamp, topical anesthesia using 0.5% tetracaine hydrochloride eye drops (Ponti-Ofteno, Laboratorios Sophia, Jalisco, Mexico) and topical 1 mg fluorescein Sodium staining (Bio-Glo, Hub Pharmaceuticals, Rancho Cucamonga CA). Post sham laser care treatment included topical eyedrops of 0.3% tobramycin and 0.1% dexamethasone (Trazidex, Laboratorios Sophia) three times daily, and 0.5 carboxymethylcellulose lubricating eye drops (Refresh-Tears, Allergan, Irving, California, USA). Topical antibiotics and corticosteroids were tapered and discontinued after two weeks.
  Interventions: Drug: Medical Treatment
- Argon Laser Treatment: Argon laser therapies were performed on an outpatient basis only by one ophthalmologist. Under slit lamp, topical anesthesia using 0.5% tetracaine hydrochloride eye drops (Ponti-Ofteno, Laboratorios Sophia, Jalisco, Mex) and topical 1 mg fluorescein Sodium staining (Bio-Glo, Hub Pharmaceuticals, Rancho Cucamonga CA) was applied. Argon laser was applied along the vessels of the pterygium apex with power between 450mW to 780 mW, spot size of 100 u with 10 milliseconds duration. Additional grill pattern treatment was given to pterygium body using a 200 microns spot size. Treatments were given in one only session. Post laser care treatment included topical eyedrops of 0.3% tobramycin and 0.1% dexamethasone (Trazidex, Laboratorios Sophia) three times daily, and 0.5 carboxymethylcellulose lubricating eye drops (Refresh-Tears, Allergan, Irving, CA, USA). Topical antibiotics and corticosteroids were tapered and discontinued after two weeks.
  Interventions: Drug: Medical Treatment; Procedure: Argon laser treatment

INTERVENTIONS:
Drug: Bevacizumab
  Other Names: Avastin
  Groups: Bevacizumab injection
Drug: Medical Treatment — Care treatment included topical eyedrops of 0.3% tobramycin and 0.1% dexamethasone (Trazidex, Laboratorios Sophia) three times daily, and 0.5 carboxymethylcellulose lubricating eye drops (Refresh-Tears, Allergan, Irving, California, USA). Topical antibiotics and corticosteroids were tapered and discontinued after two weeks.
  Groups: Medical Treatment
Drug: Medical Treatment — Care treatment included topical eyedrops of 0.3% tobramycin and 0.1% dexamethasone (Trazidex, Laboratorios Sophia) three times daily, and 0.5 carboxymethylcellulose lubricating eye drops (Refresh-Tears, Allergan, Irving, California, USA). Topical antibiotics and corticosteroids were tapered and discontinued after two weeks.
  Groups: Argon Laser Treatment
Procedure: Argon laser treatment
  Groups: Argon Laser Treatment

SUMMARY:
Blockade of vascular endothelial growth factor (VEGF) with bevacizumab has been used to treat abnormal vascular conditions of the anterior segment of the eye. In pterygium, anti-VEGF agents have been recently proposed as primary treatments, such as perioperative adjuvants, as well as treatments for pterygia recurrences after surgery. The aim of the present study was to prospectively evaluate the effect of three subconjunctival bevacizumab injections in patients with an early pterygium recurrence. Materials and Methods: The current study was a non-randomized single central trial. The method of ensuring allocation concealment was sequentially numbered. Patients with an early pterygium recurrence were selected and invited to participate in the study. Recurrence was defined as the presence of corneal vessels with concomitant conjunctival hyperemia within the first trimester after primary pterygium removal, and only patients with primary pterygium recurrence were included. Patient related factors such as pregnancy, women seeking to become pregnant, and lactating women were excluded from the study. All patients received three subconjunctival bevacizumab (2.5 mg/0.05 ml) injections (basal, 2 and 4 weeks) in the recurrence area of the pterygium, and were photographed at the third, sixth and twelfth months after the last bevacizumab injection. Photographic analyses were performed taking into account two pterygium areas: the first measure included only the vessel area in the corneal surface, while the second measure included, both, conjunctival and corneal vessel area (corneal-conjunctival area of hyperemia). Neovascularization area of each pterygium was determined using digital slit lam pictures, which were analyzed using Photoshop CS4, in order to get pixels measurements of the lesion.

DETAILED DESCRIPTION:
The method of ensuring allocation concealment was sequentially numbered. Patients with an early pterygium recurrence were selected and invited to participate in the study. Recurrence was defined as the presence of corneal vessels with concomitant conjunctival hyperemia within the first trimester after primary pterygium removal, and only patients with primary pterygium recurrence were included. Patient related factors such as pregnancy, women seeking to become pregnant, and lactating women were excluded from the study. All patients received three subconjunctival bevacizumab (2.5 mg/0.05 ml) injections (basal, 2 and 4 weeks) in the recurrence area of the pterygium, and were photographed at the third, sixth and twelfth months after the last bevacizumab injection. Photographic analyses were performed taking into account two pterygium areas: the first measure included only the vessel area in the corneal surface, while the second measure included, both, conjunctival and corneal vessel area (corneal-conjunctival area of hyperemia). Neovascularization area of each pterygium was determined using digital slit lam pictures, which were analyzed using Photoshop CS4, in order to get pixels measurements of the lesion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an early pterygium recurrence were selected and invited to participate in the study. Recurrence was defined as the presence of corneal vessels with concomitant conjunctival hyperemia within the first trimester after primary pterygium removal, and only patients with primary pterygium recurrence were included

Exclusion Criteria:

* Patient related factors such as pregnancy, women seeking to become pregnant, and lactating women. Patients with diabetes Mellitus and colagenopathies.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Patients with an early pterygium recurrence were selected and invited to participate in the study. Recurrence was defined as the presence of corneal vessels with concomitant conjunctival hyperemia within the first trimester after primary pterygium removal, and only patients with primary pterygium recurrence were included
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2012-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Pterygium recurrence | One year
  Evidence of vessel growth on both, corneal and conjunctival area after bevacizumab treatment

SECONDARY OUTCOMES:
Pterygia measurements | One year
  Measurements were performed according to Welch et al. modified technique as following: the distance in millimeters from the limbus to the apex of the lesion on the cornea (horizontal length) was performed using the slit-lamp beam (BQ 900, Haag-Streit, Koeniz, Switzerland). A standard magnification of 16 was used and the variable aperture was focused from the limbus to the apex.

OTHER OUTCOMES:
Symptoms evaluation | One year
  The frequency of symptoms (redness, watery eyes, itching, burning, foreign body sensation, and fluctuating vision) were evaluated according to Nava-Castañeda et al Questionnaire (2003). Symptoms were graded as follows: 0, never; 1, rarely (once a week); 2, occasionally (several times a week); 3, frequently (once a day); 4, usually (several times a day); and 5, continually (every hour of the day). In addition, the severity of these signs/sympots were scored at each visit on a scale of 0 to 3, with 0 representing the absence of the symptom, 1 mild, 2 moderate, and 3 severe. A total symptoms score, which is a measure of the overall severity of the patients,s conjunctival condition, was calculated by multiplying (for each individual symptom/condition) the numerical values corresponding to frequency and severity, and then adding the products for all symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Angel Nava-Castañeda, MD, Msc, Principal Investigator — Institute of Ophthalmology, Conde de Valenciana Foundation; Yonathan O Garfias, MD, PhD, Study Director — Institute of Ophthalmology, Conde de Valenciana Foundation
Locations (1):
- Institute of Ophthalmology, Conde de Valenciana Foundation, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Welch MN, Reilly CD, Kalwerisky K, Johnson A, Waller SG. Pterygia measurements are more accurate with anterior segment optical coherence tomography - a pilot study. Nepal J Ophthalmol. 2011 Jan-Jun;3(1):9-12. doi: 10.3126/nepjoph.v3i1.4271. PMID 21505540
- [Background] Nava-Castaneda A, Tovilla-Canales JL, Rodriguez L, Tovilla Y Pomar JL, Jones CE. Effects of lacrimal occlusion with collagen and silicone plugs on patients with conjunctivitis associated with dry eye. Cornea. 2003 Jan;22(1):10-4. doi: 10.1097/00003226-200301000-00003. PMID 12502940
- [Background] Nava-Castaneda A, Ulloa-Orozco I, Garnica-Hayashi L, Hernandez-Orgaz J, Jimenez-Martinez MC, Garfias Y. Triple subconjunctival bevacizumab injection for early corneal recurrent pterygium: one-year follow-up. J Ocul Pharmacol Ther. 2015 Mar;31(2):106-13. doi: 10.1089/jop.2014.0060. Epub 2014 Nov 4. PMID 25369364